CLINICAL TRIAL: NCT00558220
Title: Phase II Study of Intensive Induction (R-MegaCHOP/ESHAP)Followed By Intensive Consolidation (BEAM) In Treatment Of High-Risk Aggressive B-Cell Lymphomas
Brief Title: R-MegaCHOP-ESHAP-BEAM in Patients With High-Risk Aggressive B-Cell Lymphomas
Acronym: R-MCEB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Czech Lymphoma Study Group (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government); Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLSG 5_02; NR-8231/3
Record Dates: First submitted 2007-02-12; First posted 2007-11-14 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Diffuse Large B-Cell Lymphoma.; Primary Mediastinal B-Cell Lymphoma; Follicular Lymphoma Grade III
Keywords: Lymphoma, B-cell; Immunotherapy, passive; Remission induction; Autologous transplantation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Intensive induction followed by high-dose consolidation with stem cell support ± radiotherapy
  Interventions: Procedure: immunotherapy; Procedure: Induction treatment part 1; Procedure: Induction treatment part 2 with PBPC collection; Procedure: Induction treatment part 3; Procedure: Consolidation treatment part 1: HD-chemotherapy with ASCT; Radiation: Consolidation treatment part 2: Radiotherapy

INTERVENTIONS:
Procedure: immunotherapy — Given together with induction chemotherapy:
  Rituximab - 375 mg/m2 iv every 3 weeks, 4-6 doses
Procedure: Induction treatment part 1 — cyclophosphamide 3000 mg/m2 iv every 3 weeks, 3 cycles vincristin 2 mg iv every 3 weeks, 3 cycles doxorubicin 75 mg/m2 iv every 3 weeks, 3 cycles Prednisolone 300 mg/m2 divided into five days po every 3 weeks, 3 cycles pegfilgrastim 6 mg sc every 3 weeks.
  3 cycles consisting of combination treatment of above mentioned drugs are given.
Procedure: Induction treatment part 2 with PBPC collection — Starts three weeks after last cycle of Induction part 1.
  Etoposide 240 mg/m2 divided into equal doses for four days, together with methylprednisolone 2000 mg divided into equal doses for four days, together with cisplatin 100 mg/m2 divided into equal doses for four days, and together with cytarabine 2000 mg/m2 iv one dose on 4th day of treatment. Filgrastim 10-12 ug/kg from day five after start of chemotherapy untill stem cell collection.
  Peripheral blood progenitor cell collection (PBPC) is started when CD34 positive cells are >20/cubic milimeter of blood and continued untill 5 million of CD34 positive cells are collected from peripheral blood.
Procedure: Induction treatment part 3 — Part 3 of induction treatment is given approximately one week after the end of Part 2.
  Etoposide 240 mg/m2 divided into equal doses for four days, methylprednisolone 2000 mg divided into equal doses for four days, cisplatin 100 mg/m2 divided into equal doses for four days, cytarabine 2000 mg/m2 iv one dose on day 4 of chemotherapy and pegfilgrastim 6 mg on day five of chemotherapy are given twice three weeks apart.
Procedure: Consolidation treatment part 1: HD-chemotherapy with ASCT — Consolidation treatment Part 1 starts 4-8 weeks after the second cycle of Induction treatment Part 3.
  High dose chemotherapy (HD-chemotherapy) consists of:
  BCNU 300 mg/m2 is given on day 1, etoposide 800 mg/m2 divided into four equal doses is given on day 2-5, cytarabine 1600 mg/m2 divided into eight equal doses is given on day 2-5, melphalan 140 mg/m2 is given on day 6.
  On day 7, collected stem cells from peripheral blood (see Induction treatment part 1) are infused back to the patient. This is called autologous transplantation (ASCT). Filgrastim 5 ug/kg is given from day 14 (start of the chemotherapy being day 1) until neutrophil recovery.
Radiation: Consolidation treatment part 2: Radiotherapy — Radiotherapy is started given 4-8 weeks after the autologous transplantation. It is given to patients with initially bulky disease (>10 cm at diagnosis) or to patients with residual disease after Induction treatment part 1-3 and Consolidation treatment part 1. 30-40 Gy are given in 2 Gy fractions over 3-4 weeks.

SUMMARY:
The purpose of this study is to show if addition of Rituximab to intensive induction (MegaCHOP/ESHAP) and high-dose consolidation (BEAM) improves progression-free and overall survival in patients younger than 65 years with aggressive B-cell lymphoma and aaIPI 2 or 3.

DETAILED DESCRIPTION:
Previous study of Czech Lymphoma Study Group (4_2002)have shown that intensive induction (MegaCHOP - Cyclophosphamide 3 g/m2, Vincristine 2 mg, Adriamycin 75 mg/m2, Prednisone 300 mg/m2 every three weeks with G-CSF for three cycles, followed by ESHAP - Etoposide 240 mg/m2, Cisplatin 100 mg/m2, Solumedrol 2000 mg and cytarabine 2000 mg/m2 for three cycles every three weeks with G-CSF) followed by intensive consolidation (BEAM) and stem cell support improves progression-free survival in adult patients (18-65 years old) with aggressive B-cell lymphoma (namely, diffuse large B-cell lymphoma, primary mediastinal B-cell lymphoma and follicular lymphoma grade II) with aaIPI 2 and namely, with aaIPI 3. This study was aimed to find out if addition of four to six doses of Rituximab 375 mg/m2 on first day of every cycle of intensive induction further improves prognosis of these patients.

Inclusion criteria for this trial were:

* newly diagnosed aggressive B-cell lymphoma, namely diffuse large B-cell lymphoma, primary mediastinal B-cell lymphoma and follicular lymphoma grade III
* age 18-65 years
* age adjusted IPI (International Prognostic Index) score 2 or 3
* ECOG performance status 0-3
* signed informed consent

Exclusion criteria were:

* relapsed lymphoma
* previous treatment (up to one cycle of standard pretreatment - COP, CHOP or steroids was permitted and later became mandatory to decrease disease burden and/or improve the performance status of the patient)
* Burkitt lymphoma
* posttransplant lymphoproliferation
* CNS involvement
* other malignant tumor in previous history, except basalioma, skin squamocellular carcinoma or cervical carcinoma in situ
* other serious comorbidity

Primary endpoints was progression-free survival

Secondary endpoints were:

* rate of complete remission and overall response rate
* overall survival
* toxicity of the protocol, measured as grade III-IV toxicity and/or inability to finish the protocol as planned

Planned number of accrued patients was 100.

ELIGIBILITY:
Inclusion Criteria:

* Aggressive B-cell lymphoma, namely diffuse large B-cell lymphoma, primary mediastinal B-cell lymphoma, follicular lymphoma grade III
* Age 18-65 years
* Age-adjusted IPI score 2-3
* ECOG performance status 0-3
* Signed informed consent

Exclusion Criteria:

* Burkitt lymphoma
* Posttransplant lymphoproliferation
* Previous treatment (up to one cycle of standard pretreatment with COP, CHOP or steroids permitted and latter mandatory to decrease tumor burden and/or improve performance status)
* Other tumor in previous history with the exception of basalioma, squamous cell carcinoma of the skin or cervical carcinoma in situ
* Pregnancy/lactation
* CNS involvement
* Other serious comorbidities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2002-05; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 3 years

SECONDARY OUTCOMES:
Complete remission and overall response rate | One year
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pytlik Robert, M.D., Principal Investigator — 1st Department of Medicine, General University Hospital, Prague; Marek Trněný, M.D., PhD., Study Director — General University Hospital, Prague
Locations (8):
- Czechia (8):
  - University Hospital Brno-Bohunice, Brno
  - Hospital Chomutov, Chomutov
  - Hospital České Budějovice, České Budějovice
  - University Hospital Hradec Králové, Hradec Králové
  - University Hospital Královské Vinohrady, Prague
  - General University Hospital, Prague
  - University Hospital Motol, Prague
  - Hospital Ústí nad Labem, Ústí nad Labem

REFERENCES:
- See also: Official Site of the Czech Lymphoma Study Group — http://www.lymphoma.cz